CLINICAL TRIAL: NCT00070486
Title: Randomized Phase II Study of Eicosanoid Pathway Modulators and Cytotoxic Chemotherapy in Advanced Non-Small Cell Lung Cancer
Brief Title: Carboplatin and Gemcitabine Combined With Celecoxib and/or Zileuton in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30203; U10CA031946 (NIH); CALGB-30203; CDR0000334573 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: stage IV non-small cell lung cancer; adenocarcinoma of the lung; squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Celecoxib; Gemcitabine; zileuton

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gem + Carboplatin + Zileuton (Experimental)
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Drug: zileuton
- Gem + Carboplatin + celecoxib (Experimental)
  Interventions: Drug: carboplatin; Drug: celecoxib; Drug: gemcitabine hydrochloride
- Gem + carboplatin + zilueton + celecoxib (Experimental)
  Interventions: Drug: carboplatin; Drug: celecoxib; Drug: gemcitabine hydrochloride; Drug: zileuton

INTERVENTIONS:
Drug: carboplatin — given IV
Drug: celecoxib — given PO
  Arms: Gem + Carboplatin + celecoxib; Gem + carboplatin + zilueton + celecoxib
Drug: gemcitabine hydrochloride — given IV
Drug: zileuton — given PO
  Arms: Gem + Carboplatin + Zileuton; Gem + carboplatin + zilueton + celecoxib

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib and zileuton may stop the growth of tumor cells by stopping blood flow to the tumor and may block the enzymes necessary for tumor cell growth. Combining chemotherapy with celecoxib and/or zileuton may kill more tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of combining celecoxib and/or zileuton with carboplatin and gemcitabine in treating patients who have advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of carboplatin and gemcitabine with celecoxib and/or zileuton, in terms of 7-month progression-free survival, in patients with advanced non-small cell lung cancer.

Secondary

* Compare the response rate, distribution of survival, and failure-free survival time of patients treated with these regimens.
* Correlate CYFRA and serum vascular endothelial growth factor levels with response and survival of patients treated with these regimens.
* Correlate cyclo-oxygenase-2 and 5-lipoxygenase expression with survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes on days 1 and 8, carboplatin IV over 30 minutes on day 1, and oral zileuton 4 times daily on days 1-21.
* Arm II: Patients receive gemcitabine and carboplatin as in arm I and oral celecoxib twice daily on days 1-21.
* Arm III: Patients receive gemcitabine and carboplatin as in arm I, oral celecoxib as in arm II, and oral zileuton as in arm I.

In all arms, treatment repeats every 21 days for 6 courses. Patients with responding or stable disease continue courses of zileuton and/or celecoxib in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 1 year, every 2 months for 2 years, and then every 4 months for 3 years or until disease progression.

PROJECTED ACCRUAL: A total of 117 patients (39 per treatment arm) will be accrued for this study within 11-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) of 1 of the following cellular types:

  * Adenocarcinoma
  * Large cell
  * Squamous cell
  * Mixed
* Meets 1 of the following staging criteria:

  * Stage IIIB disease with malignant pleural effusion, supraclavicular node involvement, or contralateral hilar nodes

    * Stage IIIB patients eligible for Cancer and Leukemia Group B protocols of combined chemotherapy and chest irradiation are not allowed
  * Stage IV disease
* Measurable or nonmeasurable disease

  * Unidimensionally measurable lesions at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following are considered nonmeasurable disease:

    * Bone lesions
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Small lesions
* No leptomeningeal disease
* Symptomatic CNS metastases must be treated (e.g., surgery, radiotherapy, or gamma knife), neurologically stable, and off steroids

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 2.0 times upper limit of normal

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* None of the following within the past 6 months:

  * Myocardial infarction
  * Unstable angina
  * Symptomatic congestive heart failure
  * Serious uncontrolled cardiac arrhythmia
  * Cerebrovascular accident
  * Transient ischemic attack
  * Symptomatic carotid artery or peripheral vascular disease
  * Deep vein thrombosis
  * Significant thromboembolic event

Pulmonary

* No pulmonary embolism within the past 6 months

Gastrointestinal

* No history of gastrointestinal (GI) bleeding
* No history of peptic ulcer disease
* No active GI bleeding

Other

* Not pregnant or nursing
* No known hypersensitivity to aspirin, NSAIDs, or sulfonamides
* No currently active second malignancy other than nonmelanoma skin cancer

  * Patients are not considered to have a currently active malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for NSCLC

Chemotherapy

* No prior chemotherapy for NSCLC
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent chronic oral steroids

  * Concurrent episodic steroids for antiemetic purposes allowed
* No concurrent hormonal therapy
* Concurrent inhaled steroids allowed when medically indicated
* Concurrent megestrol for appetite stimulation is allowed

Radiotherapy

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy and recovered

Surgery

* See Disease Characteristics
* At least 2 weeks since prior surgery and recovered

Other

* No prior systemic treatments for NSCLC
* No other concurrent investigational therapy
* At least 1 week since prior nonsteroidal anti-inflammatory drugs (NSAIDs), including any of the following:

  * Rofecoxib
  * Choline magnesium trisalicylate
  * Ibuprofen
  * Naproxen
  * Etodolac
  * Oxaprozin
  * Diflunisal
  * Nabumetone
  * Tolmetin
  * Valdecoxib
* No concurrent NSAIDs
* No concurrent chronic aspirin

  * Concurrent aspirin no greater than 325 mg/day is allowed
* No concurrent fluconazole
* No concurrent leukotriene antagonists (e.g., zafirlukast, montelukast, or pranlukast)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-12; Primary Completion 2006-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Edelman, MD, Study Chair — University of Maryland Greenbaum Cancer Center
Locations (75):
- United States (75):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital at Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Edelman MJ, Watson D, Wang X, Morrison C, Kratzke RA, Jewell S, Hodgson L, Mauer AM, Gajra A, Masters GA, Bedor M, Vokes EE, Green MJ. Eicosanoid modulation in advanced lung cancer: cyclooxygenase-2 expression is a positive predictive factor for celecoxib + chemotherapy--Cancer and Leukemia Group B Trial 30203. J Clin Oncol. 2008 Feb 20;26(6):848-55. doi: 10.1200/JCO.2007.13.8081. PMID 18281656
- [Result] Edelman, MJ, Watson DM, Wang X, et al.: Eicosanoid modulation in advanced non-small cell lung cancer (NSCLC): CALGB 30203. [Abstract] J Clin Oncol 24 (Suppl 18): A-7025, 370s, 2006.